CLINICAL TRIAL: NCT06996496
Title: Examining the Implementation of an Educational Discussion Guide for Hypertensive Postpartum Patients
Brief Title: Better Understanding Patient Perspectives of an Educational Tool for Postpartum Hypertensive Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: CVS Health Foundation (Unknown)
Responsible Party: Principal Investigator, Ann C. Celi, MD, Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024P000730; GR0127667 (Other Grant/Funding Number: CVS Health Foundation)
Record Dates: First submitted 2025-05-20; First posted 2025-05-30 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Hypertension, Pregnancy Induced
Keywords: hypertension, pregnancy induced; patient satisfaction; maternal health; postpartum period; cardiovascular diseases; hypertension
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Patient Satisfaction; Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postpartum patients after hypertensive disorders of pregnancy exposed to an educational tool (Experimental): Postpartum patients after hypertensive disorders of pregnancy exposed to an educational tool
  Interventions: Other: Postpartum educational tool after hypertensive pregnancy
- Postpartum patients after hypertensive disorders of pregnancy not exposed to an educational tool (No Intervention): Postpartum patients after hypertensive disorders of pregnancy not exposed to an educational tool

INTERVENTIONS:
Other: Postpartum educational tool after hypertensive pregnancy — postpartum educational tool for patients having experienced a hypertensive disorder of pregnancy
  Arms: Postpartum patients after hypertensive disorders of pregnancy exposed to an educational tool

SUMMARY:
The goal of this clinical trial is to learn if an educational tool helps postpartum patients after having high blood pressure during their pregnancy. The main question it aims to answer is:

Does receiving this educational tool improve patient activation in the postpartum period?

Researchers will compare a group of postpartum patients who get the tool 0-2 weeks after delivery with patients who do not get the tool to see if there is a difference in their activation scores 4-12 weeks later.

Participants will:

Complete a survey at first contact with study staff

Complete a similar follow-up survey 4-12 weeks later

DETAILED DESCRIPTION:
Background and Significance

After hypertensive pregnancies, many birthing people are at increased risk of premature cardiovascular disease (CVD; Abalos et al., 2013). The transition period from obstetric care to primary care is a crucial point in the care continuum for teaching hypertension management and its benefits for longer-term improved outcomes in cardiovascular health (Phillips et al., 2022). With the rise of maternal cardiovascular mortality in the weeks after delivery and greater risks of chronic hypertension, hyperlipidemia, and cardiovascular disease in the months and years after a hypertensive pregnancy, there is a demand for improved programs for vulnerable, underserved populations immediately postpartum and into the "fourth trimester" (Phillips et al., 2022; Henderson et al., 2016). The Maternal Fetal Medicine Cardiometabolic Postpartum Clinic at Brigham and Women's Hospital (BWH) has identified gaps in knowledge and opportunities for better transitions of care from obstetricians to primary care providers (PCPs). Under the direction of Ann Celi, MD, the investigators plan to implement a program that will create improved healthcare delivery models that can be replicated locally, nationally, and internationally, resulting in better care for patients in the postpartum period. Through this work, key elements of care are being identified and thoughtful approaches are being considered to improve care. The investigators have developed a nationally and internationally recognized sustainable model with excellent appointment attendance and adherence for a racially and socioeconomically diverse patient population. This work includes a recent shift to a successful virtual platform for increased outreach to rural and vulnerable, underserved communities, including maternal health deserts. Additionally, a previous study by the investigator involved semi-structured stakeholder interviews (N=28) of patient perspectives on postpartum care at 12 BIDMC-affiliated prenatal care sites. Qualitative analysis identified themes related to key barriers and facilitators to the implementation of best practices for postpartum care, including a lack of patient understanding of postpartum care and recovery after a complicated pregnancy.

Therefore, the investigators have developed a patient discussion guide in partnership with key stakeholders from professional societies, patient advocacy foundations, and thought leaders to address these gaps in patient knowledge regarding their postpartum care and recovery and to empower patients to engage in positive health behaviors and with their primary care providers (PCPs) after transitioning from obstetric to primary care. In this study, the investigators aim to measure postpartum patients' self-reported knowledge, activation, and satisfaction related to their postpartum care, recovery, and education before participants review the discussion guide and 4-12 weeks after the participants received the discussion guide. The investigators will compare these patient knowledge, activation, and satisfaction outcomes to that of a control group that receives the discussion guide 4-12 weeks later at the time of re-contact. The investigators will also examine clinical outcomes in all study patients during the postpartum period, including blood pressure readings and number of OB and PCP visits attended, to understand patients' health behaviors and follow-up with healthcare providers. Lastly, the investigators aim to gather patient feedback on the discussion guide from the participants, any family or support people, and/or their clinical care team, as well as any barriers or facilitators for their postpartum care and recovery.

Building upon the insight gained in this study, the goal is to further disseminate these activities for the benefit of patients beyond the region. The overarching goal of this postpartum healthcare delivery program is to incorporate its components into the best care delivery models broadly. BWH is uniquely positioned to develop and lead this program as it aligns with the hospital's commitment to diversity, equity, and inclusion in clinical care, research, and educational programs.

Aims and Objectives

This study aims to measure knowledge retention, patient activation, and patient satisfaction after patients receive a discussion guide about postpartum care and recovery compared to a control group after a hypertensive pregnancy. The investigators hypothesize that, on average, patients who receive the discussion guide at the time of initial contact with study staff will report greater knowledge, activation, and satisfaction related to the participant's postpartum care, recovery, and education after receiving the discussion guide and compared to the control group. The investigators also hypothesize that participants who receive the discussion guide at the time of initial contact with study staff will have greater attendance at a follow-up with at least one visit to a PCP or OB and blood pressure control compared to the control group. The investigators seek to gain participant feedback on the discussion guide and barriers and facilitators for postpartum care and recovery. The investigators hypothesize that patients who receive the discussion guide at the time of initial contact with study staff will find it helpful for their postpartum care and recovery and easy to understand. The investigators also hypothesize that these patients will report positive feedback from their clinical care team and family/supports about the discussion guide.

Study Design

Patients receiving postpartum care at Brigham and Women's Hospital who consent to participate in this study will be randomized to either receive a discussion guide about postpartum care and recovery after a hypertensive pregnancy at the initial contact with study staff or in a few weeks after the participants complete a follow-up survey.

Patients who receive the discussion guide at the initial contact with study staff will receive the discussion guide after answering questions in a brief RedCap survey measuring their baseline knowledge retention and patient activation related to their postpartum care and recovery, and their satisfaction with postpartum education. The survey will also ask patients for their feedback on any barriers or facilitators they think will affect their postpartum care and recovery. Study staff will then recontact those patients starting approximately 4 weeks after the initial survey to complete a follow-up RedCap survey measuring self-reported knowledge retention and patient activation regarding postpartum care and recovery, and patient satisfaction with postpartum education. The survey will also ask patients for their feedback and that of any family, support people, or their clinical care team on the discussion guide, as well as any barriers or facilitators patients think are affecting postpartum care and recovery.

Patients who will receive the discussion guide after completing the follow-up survey will answer a brief RedCap survey measuring their baseline knowledge retention and patient activation related to their postpartum care and recovery, and their satisfaction with postpartum education. The survey will also ask patients for their feedback on any barriers or facilitators they think will affect their postpartum care and recovery. Study staff will then recontact those patients starting approximately 4 weeks after the initial survey to complete a follow-up RedCap survey measuring self-reported knowledge retention and patient activation regarding postpartum care and recovery, and patient satisfaction with postpartum education.

Study staff will access enrolled patients' electronic health records up to one year after delivery to learn about their transition from obstetric to primary care, including whether they attended at least one postpartum care visit, whether their blood pressure is controlled, and whether they can track and meet their health goals for postpartum recovery. Study staff may also contact enrolled patients up to five years after delivery to check-in about their long-term health after pregnancy.

Subject Selection

The investigators plan to recruit 150 patients for this study. Group A will be 75 patients who will receive the discussion guide at the time of initial contact with study staff. Group B will be a comparison group of 75 patients who will receive the discussion guide a few weeks later after completing their follow-up survey.

Patients will be recruited in-person by trained study staff on the Beyond Birth team and while on the BWH postpartum floors or the perinatal and postpartum clinic sites (BWH resident obstetric clinic, Brookside and Southern Jamaica Plain Health Centers). Patients eligible for this study will be identified by clinicians based on clinical parameters of hypertensive pregnancy and referred to study staff to be approached for this study, or by study staff accessing the minimum information necessary (e.g., hypertension diagnosis) to identify eligible patients from their medical chart in EPIC. A member of the patient's care team (e.g., attending physician, resident physician, physician assistant, midwife nurse, nurse, medical assistant, or population health manager) will obtain permission for patients to be approached by study staff. Patients will be approached at their delivery hospitalization or at an outpatient postpartum visit within approximately two weeks of delivery with the opportunity to participate in this study.

Subject Enrollment

Patients who meet the eligibility criteria will be approached by study staff on the BWH postpartum hospital floors or BWH perinatal and postpartum clinics (BWH resident obstetric clinic, Brookside and Southern Jamaica Plain Health Centers) within approximately two weeks of delivery. Back-up will be available by the study PI and/or co-investigators if needed. For patients from the medical practice of the investigator (BWH MFM clinic), patients will not be recruited by the PI about the opportunity to participate in this study, and will be assured that choosing whether to participate is completely voluntary and will not affect their clinical care in any way at any time. This will be done to ensure patients do not feel obligated to participate because their treating physician is an investigator in this study. Patients will go over a study fact sheet with a study staff member and have time to ask any clarifying questions, with the option to withdraw from the study at any time point. All patients can receive a copy of the study fact sheet once they have verbally consented to participate in the study. The study staff will obtain verbal consent from patients, as there is limited time to complete study procedures due to logistical constraints such as high patient volume and limited space in the outpatient clinics, and patients are often occupied in their recovery after just giving birth (e.g., breastfeeding, sleeping) and need to be checked on often by healthcare providers on the postpartum floors.

Study Procedures

When an eligible patient is identified, they will randomly be assigned to Group A or B using the randomization feature on MGB RedCap after they verbally consent to participate in the study and before they start the initial survey.

Group A: Patients will complete a RedCap survey on a secure electronic device given to them by the study staff gathering their demographics information and measuring their self-reported knowledge and patient activation related to their postpartum care and recovery, their satisfaction with postpartum education, and feedback on any barriers or facilitators patients think will affect their postpartum care and recovery. Patients will then be given a 3-page educational discussion guide about postpartum care and recovery after a hypertensive pregnancy, including written information and QR codes to relevant educational web pages (e.g., a short video on how to take blood pressure at home). The initial survey is estimated to take around 5-10 minutes to complete. Patients will then be recontacted by study staff via text message, email, phone call, and/or in person starting approximately 4 weeks after completion of the initial survey. Patients will be contacted up to 3 times each by text and email, once by a phone call if necessary, and in person at their 6-week postpartum outpatient visit with the opportunity to complete the follow-up survey. Study staff will attempt to recontact until approximately 12 weeks after completion of the initial survey. At the time of recontact, patients will complete a follow-up RedCap survey examining their self-reported knowledge retention of the information provided in the discussion guide and their postpartum care, patient activation to engage in their postpartum care, patient satisfaction with their postpartum education, and how helpful and understandable they found the discussion guide to be. The survey will also ask patients for their feedback and that of any family, support people, or their clinical care team on the discussion guide, as well as any barriers or facilitators patients think are affecting their postpartum care and recovery. Study staff will also access patients' electronic health records for up to 1 year after delivery to examine PCP visit attendance, OB visit attendance, blood pressure readings, and any additional hospital or healthcare provider visits for postpartum check-ups or health complications. Study staff may also contact patients up to 5 years after delivery to check-in about their long-term health after pregnancy. Scripts for study staff to follow when contacting patients up to 5 years after delivery will be submitted at a later date to the IRB for approval prior to re-contacting any patients in that later time period.

The following measure will be included in the RedCap survey for patients in Group A:

Demographics Questionnaire. Gathers relevant demographics information such as race, ethnicity, education level, and preferred method of contact.

Patient Knowledge Retention and Satisfaction Questionnaire. Assesses perceived knowledge of postpartum care and recovery and patient satisfaction with postpartum education before receiving the discussion guide and knowledge of postpartum care and recovery and satisfaction with postpartum education right at follow-up after receiving the discussion guide.

Patient Activation Measure (PAM-13). Assesses patient motivation and confidence to engage in their postpartum care. Two related free response questions about perceived barriers and facilitators related to postpartum care and recovery have been added after the PAM-13.

Group B: Patients will complete a RedCap survey on a secure electronic device given to them by the study staff gathering their demographics information and measuring knowledge and patient activation related to postpartum care and recovery, patient satisfaction with postpartum education, and feedback on any barriers or facilitators patients think will affect their postpartum care and recovery. This survey is estimated to take around 5-10 minutes to complete. Patients will then be recontacted by study staff via text message, email, phone call, and/or in person starting approximately 4 weeks after completion of the initial survey. Patients will be contacted up to 3 times each by text and email, once by a phone call if necessary, and in person at their 6-week postpartum outpatient visit with the opportunity to complete the follow-up survey. Study staff will attempt to recontact until approximately 12 weeks after completion of the initial survey. At the time of recontact, patients will complete a follow-up RedCap survey examining knowledge of and patient activation regarding their postpartum care, as well as patient satisfaction with postpartum education. The survey will also ask patients for their brief written feedback on any barriers or facilitators they think are affecting their postpartum care and recovery. Patients will then receive a copy of the discussion guide after completion of the follow-up survey through their preferred method of email, text message, in-person, or mail. Study staff will also access patients' electronic health records for up to 1 year after delivery to examine PCP visit attendance, OB visit attendance, blood pressure readings, and any additional hospital or healthcare provider visits for postpartum check-ups or health complications. Study staff may also contact patients up to 5 years after delivery to check-in about their long-term health after pregnancy. Scripts for study staff to follow when contacting patients up to 5 years after delivery will be submitted at a later date to the IRB for approval prior to re-contacting any patients in that later time period.

The following measure will be included in the RedCap survey for patients in Group B:

Demographics Questionnaire. Gathers relevant demographics information such as race, ethnicity, education level, and preferred method of contact.

Patient Knowledge Retention and Satisfaction Measure. Assesses perceived knowledge of postpartum care and recovery and patient satisfaction with postpartum education at initial approach and at follow-up.

Patient Activation Measure (PAM-13). Assesses patient motivation and confidence to engage in their postpartum care. Two related free response questions about perceived barriers and facilitators related to postpartum care and recovery have been added after the PAM-13.

ELIGIBILITY:
Patient Inclusion criteria:

* clinical diagnosis of a hypertensive disorder of pregnancy, defined as having blood pressure reading greater than 130/80
* be postpartum
* 18 or older at the time of enrollment
* able to speak, read, and understand English or Spanish.

Patient Exclusion criteria:

* no clinical diagnosis of hypertension before, during, or after their pregnancy defined as having blood pressure reading greater than 130/80
* under the age of 18
* only able to speak and read in a language other than English or Spanish
* unable to legally consent to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
patient activation measure | From enrollment to 4-12 weeks after initial contact
  Patient Activation Measure (PAM)-13 questionnaire. Range is 0-100, with higher scores representing higher patient activation.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Celi, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
This is a fundamentally a quality improvement initiative to improve iterative changes to an educational tool

REFERENCES:
- See also: link to educational tool being studied — https://www.preeclampsia.org/public/frontend/assets/img/gallery/pdf/My_Health_Beyond_Pregnancy_FINAL_2024.pdf